CLINICAL TRIAL: NCT03020589
Title: Study of Pharmacogenomic-Guided Tacrolimus Dosing and Monitoring in Kidney Transplant Recipients
Acronym: TAC3A5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-2073
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2022-07

CONDITIONS: Renal Transplant
Keywords: Renal Transplant; Tacrolimus; UNC; Phase IV
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CYP3A5 based tacrolimus dosing (Experimental): Subjects in this treatment arm will receive initial tacrolimus based on their genotype i.e., CYP3A5*1/*1 and CYP3A5*1/*3 (Expressers) will receive the initial tacrolimus dose of 0.2 mg/kg/day, with maximum of 20 mg/day in 2 divided doses. For CYP3A5*3/*3 (Non-Expressers), the subjects will receive initial tacrolimus dose of 0.1 mg/kg/day in 2 divided doses.
  Interventions: Drug: Tacrolimus
- Control (No Intervention): Subjects in the prospective control group will receive standard tacrolimus dosing as recommended per package insert and will not be dosed based on their genotype. Similarly, subjects that underwent renal transplant after 2010 and received standard tacrolimus dosing (per package insert) will serve as historical controls.

INTERVENTIONS:
Drug: Tacrolimus — See description in arm/group sections
  Other Names: Prograf, Advagraf
  Arms: CYP3A5 based tacrolimus dosing

SUMMARY:
Objective: Investigate the direct correlation of CYP3A5 genotype with tacrolimus trough levels and clinical outcomes. The primary endpoint of this study is to evaluate the proportion of patients reaching target levels (8-10 ng/mL) on Day 3 and Day 7 after kidney transplantation.

DETAILED DESCRIPTION:
Participants: All new kidney transplant recipients aged 18 to 65 years who are admitted at UNC-CH and provided informed consent will be included in this study (Unless they meet the exclusion criteria specified). A total of an anticipated 260 subjects will be included in the study, 130 of which will be included in the pharmacogenomic group and the remaining 130 will be in the control group.

Procedures (methods): The pharmacogenomic group will partake in a 12-month study comprising of two periods, Genotype-Guided Initial Dosing Intervention and Follow-up.

Briefly, patients on transplant waitlist will be screened for eligibility. At the pre-intervention assessment (Study Day 0), buccal swab samples for genotyping will be collected on all eligible patients who provided informed consent (performed in real time). Results of the genotyping test will be incorporated into electronic medical record (EMR). The initial tacrolimus dose will be based on genotype: 0.1 mg/kg/day (non- expressers) or 0.2 mg/kg/day, with maximum of 20 mg/day (expressers) given in 2 divided doses. Eligible patients who consented to receive genotype-guided tacrolimus dose will enter the pharmacogenomic group and will receive the initial tacrolimus dosing based on genotype results following kidney transplantation (Study Day 1). Subsequent tacrolimus dosing will then be adjusted according to trough concentrations (C0) and therapeutic target concentrations. The genotype-guided dosing recommendation for tacrolimus only refers to the initial tacrolimus dose. All patients in the pharmacogenomic group will be followed from Study Day 2 and up to 12 months to assess long-term outcome.

Age-, race-, and disease-matched patients who had previously received kidney transplantation with standard tacrolimus dosing from 2010 to present will also be asked to give consent for genotyping (historical controls). These patients will be included in the control group and their safety and efficacy data will be collected retrospectively for up to 12 months from the initiation of first tacrolimus dose.

As there are confounding variables, including age, race and disease state that may impact the results of the study, our study design incorporates an overall matching strategy, so that we can identify a well-matched control group. First, to control for differences in care over time, patients in the pharmacogenomic group will be matched to controls enrolled from 2010 to present. This time period was selected as there had been no major changes in standard of care or treatment regimen since 2010. After eligibility is met, control patients will be selected to match the pharmacogenomic group using a computerized matching algorithm that has been optimized to match baseline demographic and disease characteristics that have been identified a priori as likely to influence the treatment response to tacrolimus. To balance the trade-off between minimizing bias and maximizing matched sample size, a systematic approach will be conducted to identify the number of matched control patients for each patient in the pharmacogenomic group. This approach will include the following steps: 1) run the desired matching algorithm, starting with 1:1 (one control to one patient in the pharmacogenomic group) matching and iterating until the maximum desired number of potential controls per treated subject is reached; 2) for each iteration, test for covariate balance; and (3) generate numeric summaries and graphical plots of the balance statistics across all iterations in order to determine the optimal number.

The selection of patients for the control group using a matching algorithm will be conducted by an independent statistician in a blinded and unbiased manner. The statistician will have no knowledge of survival outcome, other outcome data, and genotype. The algorithm will not be used to guide treatment in any way.

ELIGIBILITY:
Inclusion Criteria:

* All new kidney transplant recipients aged 18 to 65 years who are admitted at UNC-CH and provided informed consent will be included in this study.

Exclusion Criteria:

- Patients will be excluded from participating in the study to receive genotype-guided tacrolimus dosing if he/she meets any of the exclusion criteria described below.

* Recipients who did not consent to participate in the study.
* Highly sensitized patients (ie, pretransplant T or B cell flow crossmatch positive)
* Recipients of ABO incompatible kidney transplant
* Recipients with preformed donor-specific antibodies (DSA)
* Human Leukocyte Antigen (HLA) identical kidney transplant
* Recipients of non-kidney transplant
* Recipients of repeat transplant if they are on immunosuppression at the time of transplant
* Patients using medications that have known pharmacokinetic (PK) drug interaction with tacrolimus
* Patients in whom tacrolimus therapy is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Toledo, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Univeristy of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared outside the research team.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Started | 40 | 57
Completed | 40 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control | Total
Number analyzed (Participants) | 40 | 57 | 97
Age, Continuous [Median (Full Range); unit: years] | 49 [18 to 64] | 51 [18 to 64] | 51 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 17 | 32 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 21 | 31 | 52
  White | 14 | 21 | 35
  Asian | 2 | 3 | 5
  Hispanic | 2 | 2 | 4
  American Indian or Alaska Native | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 57 | 97

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Reaching Target Tacrolimus Levels (8-10 ng/mL) on Day 3 After Kidney Transplantation
Time Frame: Day 3 after transplantation
Measure: Number; unit: proportion of participants
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
proportion of participants | 0.2 | 0.14
Statistical Analysis 1: Comparison: CYP3A5 Based Tacrolimus Dosing vs Control; Test type: Superiority; p = 0.58, Fisher Exact; Risk Ratio (RR) = 1.27, 95% CI 2-sided [0.67 to 2.05]

2. Primary Outcome: Proportion of Patients Reaching Target Tacrolimus Levels (8-10 ng/mL) on Day 7 After Kidney Transplantation
Time Frame: Day 7 after transplantation
Measure: Number; unit: Proportion of participants
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
Proportion of participants | 0.29 | 0.21
Statistical Analysis 1: Comparison: CYP3A5 Based Tacrolimus Dosing vs Control; Test type: Superiority; p = 0.46, Fisher Exact; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.72 to 2.02]

3. Secondary Outcome: Number of Events of Biopsy Proven Acute Rejection (BPAR)
Description: The number of events of BPAR within the first 3 months (Days 0 through 90), 91-180, and 181-365 days after transplantation
Time Frame: first 3 months (Days 0 through 90), 91-180, and 181-365 days after transplantation
Measure: Number; unit: BPAR events
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
BPAR events
  Days 0 through 90 | 3 | 2
  Days 91-180 | 3 | 0
  Days 181-365 | 0 | 0

4. Secondary Outcome: Tacrolimus Level
Description: Time to achieve tacrolimus therapeutic range at 0 to 4 months (8-10 ng/mL)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
Days | 6.4 (5.96) | 7.87 (5.35)

5. Secondary Outcome: Mean Number of Dose Adjustments and/or Drug Alterations
Description: Mean number of dose adjustments and/or drug alteration or addition due to insufficient immunosuppression.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Adjustments
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
Adjustments | 7.86 (2.5) | 7.37 (2.7)

6. Secondary Outcome: Percent of Participants With Chronic Renal Impairment by eGFR Category
Description: Renal function will be assessed using estimated Glomerular Filtration Rate (eGFR). Creatinine clearance (CrCl) may also be calculated as a reference. Patients will be categorized as having either mild (eGFR of 60 mL/min/1.73m^2 to 89 mL/min/1.73m^2), moderate (eGFR of 30 mL/min/1.73m^2 to 59 mL/min/1.73m^2), or severe renal impairment (eGFR <30 mL/min/1.73m^2).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
percentage of participants
  Mild : Week 1 | 23 | 24
  Mild : Month12 | 53 | 46
  Moderate : Week 1 | 35 | 42
  Moderate : Month12 | 33 | 51
  Severe : Week 1 | 43 | 35
  Severe : Month12 | 13 | 3

7. Secondary Outcome: Number of Adverse Outcomes
Description: Number of adverse outcomes (i.e., graft loss, infection, and death)
Time Frame: 12 months
Measure: Number; unit: adverse outcomes
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
Number analyzed (Participants) | 40 | 57
adverse outcomes
  Graft loss | 1 | 2
  Infection | 12 | 17
  Death | 1 | 0

8. Other Pre Specified Outcome: Direct and Indirect Costs
Description: Direct and indirect cost related to treatment and management kidney transplant recipients
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the study start through Study Day 365.
Arm/Group | CYP3A5 Based Tacrolimus Dosing | Control
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/57
Serious Adverse Events (participants affected / at risk) | 4/40 | 2/57
Other Adverse Events (participants affected / at risk) | 40/40 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP3A5 Based Tacrolimus Dosing (N=40) | Control (N=57)
Biopsy Proven Acute Rejection (Renal and urinary disorders) | 4 (6) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP3A5 Based Tacrolimus Dosing (N=40) | Control (N=57)
Neurotoxicity (Nervous system disorders) | 3 (5) | 5 (5)
Tremor (Nervous system disorders) | 10 (12) | 22 (25)
Headache (Nervous system disorders) | 11 (16) | 21 (26)
Diarrhea (Gastrointestinal disorders) | 12 (16) | 22 (37)
Nausea (Gastrointestinal disorders) | 12 (26) | 21 (28)
Constipation (Gastrointestinal disorders) | 9 (18) | 9 (12)
Vomiting (Gastrointestinal disorders) | 8 (14) | 10 (15)
Hypertension (Cardiac disorders) | 11 (24) | 25 (40)
Abnormal renal function (Renal and urinary disorders) | 23 (56) | 39 (73)
Increase creatinine (Renal and urinary disorders) | 20 (36) | 21 (29)
Delayed Graft Function Requiring Dialysis (Renal and urinary disorders) | 13 (13) | 12 (12)
Leukopenia (Blood and lymphatic system disorders) | 30 (86) | 37 (101)
Anemia (Blood and lymphatic system disorders) | 39 (115) | 56 (96)
Hyperkalemia (Metabolism and nutrition disorders) | 28 (65) | 44 (90)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (89) | 23 (53)
Hypomagnesemia (Metabolism and nutrition disorders) | 33 (94) | 53 (145)
Hypophosphatemia (Metabolism and nutrition disorders) | 20 (34) | 27 (48)
Hyperlipidemia (Metabolism and nutrition disorders) | 7 (7) | 14 (16)
Edema (Metabolism and nutrition disorders) | 9 (20) | 12 (22)
Infection (Infections and infestations) | 10 (12) | 12 (17)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9) | 8 (9)
Graft loss (Renal and urinary disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03020589/Prot_SAP_000.pdf